CLINICAL TRIAL: NCT04056390
Title: Ablation STrategies for Repeat PrOcedures in Patients With Atrial Fibrillation Recurrences
Acronym: ASTRO AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Collaborators: Medtronic (Industry); CRO Kottmann (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF124/2017
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Substrate Modification (Active Comparator): After obtaining a voltage map of the LA, substrate modification by catheter ablation using an irrigated radio frequency current ablation catheter will be performed aiming at low-voltage areas (LVA) < 0.5mV.
  Interventions: Procedure: Catheter ablation using irrigated radiofrequency current ablation or cryothermal energy
- LAA Isolation (Active Comparator): Patients will undergo LAA-isolation using the cryoballoon (CB). Six weeks later patients will undergo re-mapping. In case of residual conduction LAA-reisolation will be performed. In case of durable LAA isolation, interventional LAA occlusion is recommended.
  Interventions: Procedure: Catheter ablation using irrigated radiofrequency current ablation or cryothermal energy

INTERVENTIONS:
Procedure: Catheter ablation using irrigated radiofrequency current ablation or cryothermal energy — Substrate ablation in terms of voltage abatement versus electrical left atrial appendage isolation.

SUMMARY:
The aim of the study is to evaluate different ablation strategies in patients with AF recurrences despite chronic PVI after prior catheter ablation.

The present study is a multi-centre prospective randomized study enrolling 256 patients with drug-refractory AF despite previous AF ablation.

After PV remapping confirming durable PVI patients will be assigned to 2 different groups: Group A: Substrate modification.

After obtaining a voltage map of the LA, substrate modification will be performed aiming at low-voltage areas (LVA) < 0.5mV.

Group B: LAA isolation. Patients will undergo LAA-isolation using the cryoballoon (CB). Catheter ablation procedures will be performed with commercially available devices including 3D mapping systems (CARTO, EnSite) and irrigated radiofrequency current (RFC) ablation or cryothermal balloon ablation (Arctic Front Advance).

The primary endpoint is freedom from documented recurrence of AF or any atrial tachyarrhythmia lasting > 30 seconds between day 91 and 365 after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Symptomatic non-valvular atrial fibrillation despite prior ablation with an indication for re-ablation according to current guidelines.

  * Permanent pulmonary vein isolation according to mapping with a spiral mapping catheter
  * Age 18-85 years.
  * Left atrial size < 55mm.
  * Left ventricular ejection fraction ≥ 45%.
  * Patient is able to provide informed consent and is willing to comply with the study protocol.

Exclusion Criteria:

* Contraindications for repeat ablation
* Reconnected pulmonary veins according to mapping results with a spiral mapping catheter
* Minimal diameter of LAA neck ≥25mm
* History of mitral valve surgery
* Severe mitral valve regurgitation
* Inability to be treated with oral anticoagulation
* Presence of intracardiac thrombi
* Chronic obstructive pulmonary disease treated with long acting bronchodilatators
* Asthma
* Obstructive sleep apnea syndrome
* Pregnancy
* Participation in other clinical studies
* Unwilling to follow the study protocol and to attend follow-up visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia Recurrence | Day 91-365 after index ablation
  Freedom from AF/AT

SECONDARY OUTCOMES:
Incidence of periprocedural complications | day 0 - day 365
  Incidence of periprocedural complications such as cardiac perforation, thromboembolic events or bleeding
Number of electrical cardioversions and hospitalizations | day0 - day 365
  Number of electrical cardioversions and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Boris Schmidt, MD, Principal Investigator — Cardioangiologisches Centrum Bethanien
Locations (7):
- Germany (7):
  - Klinik für Elektrophysiologie/Rhythmologie - Herz- und Diabeteszentrum NRW - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Universitätsklinikum Köln, Cologne
  - Cardioangiologisches Centrum Bethanien, Frankfurt am Main
  - Universitätsmedizin Greifswald, Greifswald
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg, Hamburg
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Universitäts Klinikum Ulm, Ulm

REFERENCES:
- [Derived] Schmidt B, Bordignon S, Metzner A, Sommer P, Steven D, Dahme T, Busch M, Tilz RR, Schaack D, Rillig A, Sohns C, Sultan A, Weinmann-Emhardt K, Hummel A, Vogler J, Fink T, Lueker J, Pott A, Heeger C, Chun KRJ. Ablation Strategies for Repeat Procedures in Atrial Fibrillation Recurrences Despite Durable Pulmonary Vein Isolation: The Prospective Randomized ASTRO AF Multicenter Trial. Circulation. 2024 Dec 17;150(25):2007-2018. doi: 10.1161/CIRCULATIONAHA.124.069993. Epub 2024 Oct 7. PMID 39371020